CLINICAL TRIAL: NCT04839588
Title: Home-based Virtual Reality System for the Treatment of Chemotherapy-related Cognitive Impairments
Brief Title: Telerehabilitation Cognitive Impairments Following Chemotherapy Usability Study
Acronym: TCIFCU
Status: Completed | Type: Observational
Sponsor: Bright Cloud International Corp (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: Telerehab CH Usability; R43CA232936 (NIH)
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Chemotherapy-Related Cognitive Impairment; Healthy
Keywords: chemotherapy; cognitive impairments; breast cancer
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Cognitive Dysfunction; Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usability study, healthy volunteers and those with cognitive impairments following chemotherapy: 2 elderly healthy volunteers and 2 participants with lasting cognitive impairments following chemotherapy for breast cancer. All will perform evaluation of a computer-based experimental system. Participants will be
  * Female Either healthy or breast cancer survivor;
  * Age 20 to 65 years;
  * Have st least 12 years of formal education;
  * Be English speakers;
  Interventions: Other: Usability study

INTERVENTIONS:
Other: Usability study — Participants will first be screened for propensity to simulation sickness and for cognitive state using the MoCA evaluation test. Those who passed the screening will perform 4 usability sessions rating the ease of use and perceived benefit of the experimental system and of a caregiver interface laptop. The 2 healthy volunteers will evaluate first, such that issues may be resolved before testing is done on the impaired participants. Each session will be compensated with a $35 payment. During each session participants will play a series of increasing difficulty simulated tasks, aimed to train primarily the executive functions domain. At the end of each session participants will rate their experience using custom subjective evaluation forms with multiple items. Each item will be scored using a 5-point Likert scale. At the end of the 4th session, participants will also fill the USE standardized usability form.
  This usability evaluation will be conducted at the NJ Bioscience Center.

SUMMARY:
Develop a game-based upper-extremity motor and cognitive rehabilitation system using custom and adaptable virtual reality simulations.

Perform usability study on 2 elderly healthy volunteers and 2 breast cancer survivors with lasting cognitive impairments following chemotherapy, so to improve the product design. The usability evaluation will be done at NJ Bioscience Center (North Brunswick, NJ).

DETAILED DESCRIPTION:
The study will generate data on ease of use of a system for subjects with stage II or stage III breast cancer survivors with lasting cognitive impairments subsequent to their first chemotherapy regimen. The usability component will uncover technical issues in its usability, as well as its rating on perceived usefulness. Data will also be collected on the ease of remote monitoring of the subjects by clinicians.

This portion of the study is intended to provide information pertaining to the usability of the experimental system for remote integrative (cognitive and motor) therapy of breast cancer survivors (Stage II or III) with lasting chemotherapy related cognitive impairment (CRCI) subsequent to first chemotherapy regimen, living in the community.

Specific aims are:

1. testing of a added biosensors, new technology acceptance and ease of use at home by these individuals;
2. a caregiver console and enhanced automatic session report that will allow remote monitoring of patient exercising and offline data processing and review.

Participants will each perform 4 usability evaluation sessions. At the end of each session participants will fill a custom evaluation form, using 5-point Likert scale scoring. At the end of the last session participants will also fill a USE standardized usability evaluation form.

ELIGIBILITY:
At NJ Bioscience Center Healthy Volunteers

* Female
* Age 20 to 65;
* Good or corrected hearing;
* Good or corrected vision;
* No motor or cognitive impairments;
* English speakers;
* Those with low propensity for simulation sickness (as determined by the Simulation Sickness Questionnaire [Kennedy et al, 1993]).
* Either healthy or having had stage II or stage III breast cancer;
* Montreal Cognitive Assessment (MoCA) Score 10-25 indicating mild to moderate impairment [Chapman 2016] or 26-30 indicating normal cognition;

EXCLUSION CRITERIA

* Male;
* Female participants younger than 20 or older than 65;
* High propensity for simulation sickness (as determined by Simulation Sickness Questionnaire screening);
* Those with severe visual neglect or legally blind;
* Those with severe hearing loss or deafness;
* Those with uncontrolled hypertension (>190/100 mmHg);
* Those with severe cognitive impairment (MoCA score<10);
* Current diagnosis of moderate-severe depression (Beck Depression Inventory II score of 17-63);
* a history of psychiatric illness, defined as serious psychiatric illness such as bipolar mood disorder and schizophrenia, or requiring psychiatric hospitalization.
* a history of or current substance abuse;
* a previous head injury resulting in loss of consciousness;
* a prior diagnosis of neurological illness;
* a current or prior diagnosis of brain cancer;
* non-English speakers;
* Those unable to reliable participate in pre-study assessment due to any reason;
* Those with co-morbidities limiting arm and neck motor function (ex. lymphedema, chronic pain, severe arthritis);
* Less than 1 month post first chemotherapy regimen or starting chemotherapy during 16 weeks post screening (as chemotherapy during study participation is a confounding factor);
* Those with Stage IV (metastatic) breast cancer will be excluded;
* Those presenting with multiple cancers, such as breast and arm bone cancer, or breast and brain cancer;
* Those who are unwilling to allow a home inspection to ascertain Internet quality, determine best placement for the experimental or sham systems, for installation and removal of the systems and necessary repairs.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the study targets breast cancer survivors, participants will all be female. Breast cancer prevalence is overwhelmingly in women.
Study Population: The targeted subjects will be either breast cancer survivors, living in the community, without requiring transfers, or healthy, age-matched volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
USE questionnaire to assess the usability of a computerized system | At the end of the 4th evaluation session (about 1 month from enrollment)
  A standardized questionnaire to assess the usefulness, satisfaction and ease of use of the experimental system [Lund, 2001] when evaluated by study participants. The form consists of 30 questions, each rated on a 7-point Likert scale (1 worst 7 best). The score range for this form is 30 (min) to 210 (max).
  Participants will also be able to comment in free form on aspects they liked most and least about the device.

SECONDARY OUTCOMES:
Subjective rating questionnaire of the device and therapy | At each of 4 evaluation sessions over 1 month from enrollment
  Participants rate the usefulness, satisfaction issues, and ease of use of the experimental system and its therapeutic games, as well as ease of use of the Caregiver laptop. The Subjective Evaluation Form consists of questions, each rated on a 5-point Likert scale (1 worst to 5 best outcome).

OTHER OUTCOMES:
Simulation Sickness Questionnaire for participant | Screening at consent (one time)
  Form used at screening post-consent to determine a participant's propensity for simulation sickness [Kennedy et al.,1993]. The questionnaire asks participants to score 16 symptoms on a four point scale (0-3). Score range is 0 (best outcome - no likelihood of experiencing simulation sickness with the device) to 48 (worst outcome - certainty that the participant will experience severe simulation sickness).
Cyber-sickness Susceptibility Questionnaire for participant | Screening at consent (one time)
  Form used at screening post-consent to determine a participant's propensity for simulation sickness [Freiwald et al., 2020]. The questionnaire asks participants 26 questions The first 13 questions ascertain the general heath and fitness of the subject, and have Yes/No answers The remaining 13 questions are score on a on a 5 point Likert scale, with five point Likert scales, referring to the frequency of each complaint's occurrence. These scales range from 0 to 4 with the labels "very rarely", "rarely", "occasionally", "frequently" and "very often".
Montreal Cognitive Assessment (MoCA) to measure level of cognitive impairment | Screening at consent (one time)
  Used at screening post-consent to determine level of cognitive impairment [Nasreddine et al 2005] for participants. The form has a score range from 0 (worst) to 30 (best) - no cognitive impairments. For the participants with early Alzheimer's Disease the form will confirm the participant is in the score range of 19-25.
Biosensor readings | At each of 4 evaluation sessions over 1 month from enrollment
  Custom biosensors will provide additional data which will be used to gauge levels of cognitive engagement with the tasks performed during the evaluation.
Game difficulty level | At each of 4 evaluation sessions over 1 month from enrollment
  Game difficulty level when performing a simulated game task using the experimental system. Levels are 1 (easiest) to 16 (hardest)
Heart rate | Before and after each of 4 evaluation sessions over 1 month from enrollment
  Heart rate (Pulse) measured with a medical meter at start and end of each usability evaluation session
Blood pressure (systolic and diastolic) | Before and after each of 4 evaluation sessions over 1 month from enrollment
  Blood pressure (Systolic and diastolic) measured with a medical meter before and after each Usability evaluation session.

CONTACTS AND LOCATIONS:
Overall Officials: Grigore C Burdea, PhD, Principal Investigator — Bright Cloud Int'l Corp
Locations (2):
- United States (2):
  - Bright Cloud Int'l Corp, North Brunswick, New Jersey
  - New Jersey Bioscience Center, North Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No
We will not disclose data on individual participants.

REFERENCES:
- See also: Description: BCI's corporate site showing therapeutic games used with the device — http://www.BrightBrainer.com